CLINICAL TRIAL: NCT01196598
Title: Impact of Pelvic Floor Muscle Training and Hypopressive Exercises in Women With Pelvic Organ Prolapse: Randomized Controlled Trial
Brief Title: Pelvic Floor Muscle Training and Hypopressive Exercises for Pelvic Organ Prolapse
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Ana Paula Magalhães Resende, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1978/07
Record Dates: First submitted 2010-09-01; First posted 2010-09-08 (Estimated); Last update posted 2010-09-08 (Estimated); Status verified 2010-08

CONDITIONS: Pelvic Organ Prolapse
Keywords: pelvic floor; pelvic organ prolapse
MeSH Terms: conditions — Pelvic Organ Prolapse | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PFMT group (Active Comparator): Women who undergo to three months of a pelvic floor muscle training program.
  Interventions: Other: Exercises
- HE + PFM group (Active Comparator): Women who undergo to three months of a hypopressive exercises plus pelvic floor muscle contraction program.
  Interventions: Other: Exercises
- HE group (Active Comparator): Women who undergo to three months of a hypopressive exercises program.
  Interventions: Other: Exercises
- Control (Active Comparator): Women who undergo to a session for lifestyle advice.
  Interventions: Other: Exercises

INTERVENTIONS:
Other: Exercises — Three individual initial sessions for learn about pelvic floor muscle localization and function; receive lifestyle advice and practice the exercises correctly.
  The control group receive only lifestyle advice.
  Followed by three months of home training with appointments each two weeks with physiotherapist.

SUMMARY:
To verify if pelvic floor muscle training program and/or a hypopressive exercise program could improve women with stage II of pelvic organ prolapse, their symptoms or pelvic floor muscle strength.

DETAILED DESCRIPTION:
To verify if three months of an exercise program could improve stage II of pelvic organ prolapse, as a conservative treatment.

ELIGIBILITY:
Inclusion Criteria:

* women with stage II of pelvic organ prolapse, preferably symptomatic and not to be submitted to surgery to correct pelvic organ prolapse during the study

Exclusion Criteria:

* Neuromuscular diseases and use of hormonal therapy

Ages: 40 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2008-01; Primary Completion 2010-10 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Pelvic floor muscle changes | 3 months after the begining of treatment
  Digital palpation - Evaluates the pelvic floor muscle contraction and assign values according to scales: Oxford (previously validated) and muscular endurance (measured in seconds)
  Surface electromyography - evaluates the electrical activity generated by activation of motor units of pelvic floor muscles - during the rest and during the maximum voluntary contraction
  2D perineal ultrasound - evaluates the cross sectional area of levator ani muscle.

SECONDARY OUTCOMES:
Pelvic Organ Prolapse changes | 3 months after the begining of treatment
  Quantification of stage of pelvic organ prolapse. Measured during gynecology exam by pelvic organ prolapse quantification (POP-Q)exam.
  Measure of changes in symptoms of pelvic organ prolapse using a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Ana Paula M. Resende, Principal Investigator — Post graduate student
Locations (1):
- Federal University of São Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Resende APM, Bernardes BT, Stupp L, Oliveira E, Castro RA, Girao MJBC, Sartori MGF. Pelvic floor muscle training is better than hypopressive exercises in pelvic organ prolapse treatment: An assessor-blinded randomized controlled trial. Neurourol Urodyn. 2019 Jan;38(1):171-179. doi: 10.1002/nau.23819. Epub 2018 Oct 12. PMID 30311680
- [Derived] Bernardes BT, Resende AP, Stupp L, Oliveira E, Castro RA, Bella ZI, Girao MJ, Sartori MG. Efficacy of pelvic floor muscle training and hypopressive exercises for treating pelvic organ prolapse in women: randomized controlled trial. Sao Paulo Med J. 2012;130(1):5-9. doi: 10.1590/s1516-31802012000100002. PMID 22344353